CLINICAL TRIAL: NCT06329557
Title: Optimizing the Patient Experience Through Provider Coaching or Communication Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Summer V. Allen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-007188
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Patient Satisfaction; Communication
MeSH Terms: conditions — Patient Satisfaction; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Survey and Coaching (Active Comparator): Individual coaching with a trained patient experience professional (XTEC coach) will occur individually with clinicians 3-4 times over several weeks. The coach will assist participants with improving communication with patients.
  Interventions: Behavioral: Intervention 1
- Survey and Communication Class (Active Comparator): A one-hour communication class will take place during the workday. The class will be offered virtually or in person for a group of clinicians to attend.
  Interventions: Behavioral: Intervention 1
- No Intervention (No Intervention): Surveys only

INTERVENTIONS:
Behavioral: Intervention 1 — Intervention 3
  Other Names: Intervention 2
  Arms: Survey and Coaching; Survey and Communication Class

SUMMARY:
Hypothesis: Clinicians who receive patient experience coaching or communication classes have improved patient satisfaction scores and improved clinician satisfaction.

DETAILED DESCRIPTION:
Aims, purpose, or objectives:

To identify if patient experience coaching or communication classes have an effect on patient satisfaction scores and clinician satisfaction.

ELIGIBILITY:
Inclusion Criteria:

• Clinicians of Primary Care Mayo Clinic

Exclusion Criteria:

* Not clinicians of Primary Care Mayo Clinic or Residents within Rochester Primary Care Clinicians from Family Medicine, or Clinicians from Community Internal Medicine Geriatrics, Palliative Medicine, and Community Pediatrics and Adolescent Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To identify if patient experience coaching or communication classes have an effect on patient satisfaction scores and clinician satisfaction. | 1 year
  Participants will be sent a Pre-test Questionnaire and Maslach Burnout Inventory within the introductory email containing a RedCap link for them to use if they desire to participate. Immediately following the intervention, and two months after the intervention, participants will receive a Maslach Burnout Inventory to complete.
  Method used:
  Average Emotional Exhaustion- Higher the scores indicate higher degree of burnout Depersonalization- Higher scores indicate higher degree of burnout Personal Accomplishment- Lower scores indicate higher degree of burnout

CONTACTS AND LOCATIONS:
Overall Officials: Summer V Allen, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota